CLINICAL TRIAL: NCT02748252
Title: Prognosis of a First-Ever Stroke in Persons Living With HIV
Acronym: PROFES
Status: Terminated | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AMR_2014-3
Record Dates: First submitted 2016-04-18; First posted 2016-04-22 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Cerebrovascular Accident, Acute; HIV
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV patients: HIV patients admitted in Stroke units for the first occurence of acute stroke
  Interventions: Other: stroke center referral
- non HIV patients: non HIV patients admitted in Stroke units for the first occurence of acute stroke
  Interventions: Other: stroke center referral

INTERVENTIONS:
Other: stroke center referral

SUMMARY:
With aging of the persons living with HIV, cardiovascular diseases now account for substantial mortality and morbidity. Stroke frequency grows exponentially with aging and its incidence doubles every decade over 55 years of age.

The prognosis of ischemic stroke depends mainly on the care in Stroke Units in the acute phase of the disease (thrombolysis/thrombectomy). It is important that HIV patients are referred to these units in the first hours of a stroke and not to their infectious disease units which is a loss of chance.

It would also be important to know whether HIV patients need specific protocols for stroke emergency management.

The study aims to compare the functional prognosis after the first occurrence of an ischemic stroke, in patients admitted to a Stroke Unit, whether they are infected or not infected by HIV.

ELIGIBILITY:
Inclusion Criteria:

* Patients unexposed to HIV: HIV-1 seronegative OR patients exposed to HIV: HIV seropositive for over 6 months with or without antiretroviral treatment. Confirmed by Elisa and Western blot tests
* admitted for ischemic stroke, defined as a sudden cerebrovascular event confirmed by MRI
* at least 18 years of age
* paired with patients unexposed to HIV, admitted for ischemic stroke, same gender and age

Exclusion Criteria:

* antecedents of a symptomatic ischemic or hemorrhagic cerebrovascular event
* no social security benefits;
* Absence of signed informed consent for the study
* Patients currently pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to a Stroke Unit for the first occurrence of an ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
degree of disability measured with the modified Rankin Scale | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris, France

IPD SHARING:
Plan to Share IPD: No